CLINICAL TRIAL: NCT07215481
Title: Quantitative Digitography to Evaluate the Efficacy of Image Guided Algorithmic DBS Programming
Brief Title: Automated Image-Guided Programming of Deep Brain Stimulation (DBS) for Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Helen M. Bronte-Stewart, Professor of Neurology and Neurological Sciences, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 83174
Record Dates: First submitted 2025-10-09; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Parkinson's Disease (PD)
Keywords: deep brain stimulation; DBS; PD; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Deep Brain Stimulation (Experimental): Participants start with a sham condition (baseline) for approximately 45 minutes. Participants then receive the following four deep brain stimulation conditions in a randomized order for approximately 45 minutes each delivered by the Boston Scientific Vercise Genus neurostimulator. Neither the participants nor the assessor will be aware of what condition they receive. Before starting the condition, there will be a wash in for approximately 15 minutes. Participants will then perform tasks and questionnaires for approximately 30 minutes on each condition.
  The four conditions are:
  1. Standard of Care Deep Brain Stimulation
  2. Illumina 3D Deep Brain Stimulation
  3. Illumina 3D Deep Brain Stimulation Reduced Amplitude
  4. Illumina 3D Deep Brain Stimulation Higher Amplitude
  Interventions: Device: Shame Control (Baseline); Device: Standard of Care Deep Brain Stimulation; Device: Illumina 3D Deep Brain Stimulation; Device: Illumina 3D Deep Brain Stimulation Reduced Amplitude; Device: Illumina 3D Deep Brain Stimulation Higher Amplitude

INTERVENTIONS:
Device: Shame Control (Baseline) — Participant's device (Boston Scientific Vercise Genus neurostimulator) is turned off for 45 minutes.
Device: Standard of Care Deep Brain Stimulation — Participant's device (Boston Scientific Vercise Genus neurostimulator) is turned 'ON' for 45 minutes using a configuration and amplitude determined as standard of care by the clinician.
Device: Illumina 3D Deep Brain Stimulation — Participant's device (Boston Scientific Vercise Genus neurostimulator) is turned 'ON' for 45 minutes using a configuration and amplitude determined by the automated Illumina 3D algorithm.
Device: Illumina 3D Deep Brain Stimulation Reduced Amplitude — Participant's device (Boston Scientific Vercise Genus neurostimulator) is turned 'ON' for 45 minutes using a configuration and amplitude determined by the automated Illumina 3D algorithm but at a reduced stimulation amplitude.
Device: Illumina 3D Deep Brain Stimulation Higher Amplitude — Participant's device (Boston Scientific Vercise Genus neurostimulator) is turned 'ON' for 45 minutes using a configuration and amplitude determined by the automated Illumina 3D algorithm but at a higher stimulation amplitude.

SUMMARY:
The goal of this clinical trial is to evaluate an automated deep brain stimulation (DBS) algorithm developed by Boston Scientific called Illumina 3D for motor symptoms in Parkinson's disease (PD). The main question it aims to answer is: Is this new automated algorithm effective for treating motor symptoms of PD. Fifteen participants are anticipated to be enrolled.

Participants are individuals who recently were implanted with DBS in the subthalamic nucleus as part of their regular clinical treatment and are scheduled to have their DBS turned ON for the first time. In addition to their regular clinical visit when their DBS is turned ON by their clinician, participants are tested on DBS settings determined by Illumina 3D (an automated algorithm). Participants are tested on these different settings across different motor tasks, including walking and finger tapping, as well as answering questionnaires. The experiment is expected to last 1 or 2 days; this is not a longitudinal or long-term trial. Participants return to their usual DBS settings once they leave the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease (PD)
* Newly implanted or soon to be implanted with deep brain stimulation (Boston Scientific device)
* Willingness to withdraw from clinical medication regimen when necessary for research visits

Exclusion Criteria:

* Dementia
* Unable or unwilling to come OFF DBS for a short period of time

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in QDG Mobility Score (OFF DBS to Illumina 3D) | Baseline and after 45 minutes of Illumina 3D DBS
  Quantitative Digitography (QDG) Mobility Score is a single score representing a participant's overall movement proficiency by combining performance across different aspects of movement including speed, frequency, amplitude, and rhythmicity measured using an engineered Keyduo QDG device during an alternating finger pressing and releasing with the index and middle finger. It is represented by a single value between 0 and 100 for each hand, where 100 represents ideal performance. The primary outcome is the difference in QDG Mobility Score from the OFF DBS condition (baseline) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG mobility score will be used.

SECONDARY OUTCOMES:
Change in QDG Tremor Severity Score (OFF DBS to Illumina 3D) | Baseline (OFF DBS) and after 45 minutes of Illumina 3D DBS
  A single score representing the proportion and amplitude of tremor-identified strikes using an engineered Keyduo QDG device. It is represented by a single value between 0 and 100, where 100 represents the worst tremor severity. A secondary outcome is the difference in QDG Tremor Severity Score from the OFF DBS condition (Baseline) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in QDG Percent Rest Tremor (OFF DBS to Illumina 3D) | Baseline (OFF DBS) and after 45 minutes of Illumina 3D DBS
  The proportion of tremor-identified strikes using an engineered Keyduo QDG device. Range from 0 to 100%. A secondary outcome is the difference in QDG Percent Rest Trremor from the OFF DBS condition (Baseline) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in QDG Press Amplitude (OFF DBS to Illumina 3D) | Baseline (OFF DBS) and after 45 minutes of Illumina 3D DBS
  The average amplitude of strikes using an engineered Keyduo QDG device. Ranges from 0 to 14 mm. A secondary outcome is the difference in QDG Press Amplitude from the OFF DBS condition (Baseline) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in QDG Press Amplitude Coefficient of Variation (OFF DBS to Illumina 3D) | Baseline (OFF DBS) and after 45 minutes of Illumina 3D DBS
  The coefficient of variation of press amplitude of strikes using an engineered Keyduo QDG device. A secondary outcome is the difference in QDG Press Amplitude Coefficient of Variation from the OFF DBS condition (Baseline) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in QDG Interstrike Interval (OFF DBS to Illumina 3D) | Baseline (OFF DBS) and after 45 minutes of Illumina 3D DBS
  The interstrike-interval (i.e., the time it takes to complete one full press and release of the lever) of alternating tapping will be measured using an engineered Keyduo QDG device. The interstrike-interval is a time in milliseconds. A secondary outcome is the difference in QDG Interstrike Interval from the OFF DBS condition (Baseline) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in QDG Release Slope (OFF DBS to Illumina 3D). | Baseline (OFF DBS) and after 45 minutes of Illumina 3D DBS
  The average speed of release using an engineered Keyduo QDG device. Units of cm/s. A secondary outcome is the difference in QDG Release Slope from the OFF DBS condition (Baseline) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in QDG Press Speed (OFF DBS to Illumina 3D) | Baseline (OFF DBS) and after 45 minutes of Illumina 3D DBS
  The average speed of the press using an engineered Keyduo QDG device. Units of cm/s. A secondary outcome is the difference in QDG Press Speed from the OFF DBS condition (Baseline) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in QDG Interstrike Interval Coefficient of Variation (OFF DBS to Illumina 3D) | Baseline (OFF DBS) and after 45 minutes of Illumina 3D DBS
  The variability of the interstrike-interval of alternating tapping, as quantified by the coefficient of variation, will be measured using an engineered Keyduo QDG device. A secondary outcome is the difference in QDG Interstrike interval coefficient of varation from the OFF DBS condition (Baseline) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in QDG Percent Freezing (OFF DBS to Illumina 3D) | Baseline (OFF DBS) and after 45 minutes of Illumina 3D DBS
  Proportion of freezing of finger tapping using a validated algorithm. Range from 0 to 100%. A secondary outcome is the difference in QDG Percent Freezing from the OFF DBS condition (Baseline) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in Gait Speed (OFF DBS to Illumina 3D) | Baseline (OFF DBS) and after 45 minutes of Illumina 3D DBS
  The time it takes a person to walk a specified distance on level ground as measured by the GaitRite. Reported as m/s. A secondary outcome is the difference in gait speed from the OFF DBS condition (Baseline) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in Gait Arrhythmicity (OFF DBS to Illumina 3D) | Baseline (OFF DBS) and after 45 minutes of Illumina 3D DBS
  Stride (gait cycle) time will be measured using the GaitRite. Gait arrhythmicity is defined as the mean stride time coefficient of variation (CV) of both legs. A greater stride time CV is indicative of less rhythmic gait/stepping. A secondary outcome is the difference in gait arrhythmicity from the OFF DBS condition (Baseline) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in MDS-UPDRS III Total Score (OFF DBS to Illumina 3D) | Baseline (OFF DBS) and after 45 minutes of Illumina 3D DBS
  PD symptoms will be assessed clinically using the MDS-Unified Parkinson's Disease Rating Scale (UPDRS) Section III. This is a motor examination to evaluate speech, facial expression, tremor at rest, action or postural tremor of hands, rigidity, finger taps, hand movements, rapid alternating movement of hands, leg agility, arising from chair, posture, gait, freezing of gait, posture, body bradykinesia, and postural stability. Each item is scored on a scale from 0 (normal) to 4 (severe), with the total possible score ranging from 0 to 132. A secondary outcome is the difference in MDS-UPDRS III from the OFF DBS condition (Baseline) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in MDS-UPDRS III Bradykinesia Subscore (OFF DBS to Illumina 3D) | Baseline (OFF DBS) and after 45 minutes of Illumina 3D DBS
  Bradykinesia-related items of the MDS-UPDRS III, which includes items 3.4-3.8. Each item is scored on a scale from 0 (normal) to 4 (severe), with the total possible score ranging from 0 to 40. A secondary outcome is the difference in MDS-UPDRS III Bradykinesia subscore from the OFF DBS condition (Baseline) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in MDS-UPDRS III Rigidity Subscore (OFF DBS to Illumina 3D | Baseline (OFF DBS) and after 45 minutes of Illumina 3D DBS
  Rigidity-related items of the MDS-UPDRS III, which includes item 3.3. Each item is scored on a scale from 0 (normal) to 4 (severe), with the total possible score ranging from 0 to 20. A secondary outcome is the difference in MDS-UPDRS III Rigidity subscore from the OFF DBS condition (Baseline) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in MDS-UPDRS III Tremor Subscore (OFF DBS to Illumina 3D) | Baseline (OFF DBS) and after 45 minutes of Illumina 3D DBS
  Tremor-related items of the MDS-UPDRS III, which includes items 3.15-3.18. Each item is scored on a scale from 0 (normal) to 4 (severe), with the total possible score ranging from 0 to 40. A secondary outcome is the difference in MDS-UPDRS III Tremor subscore from the OFF DBS condition (Baseline) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in MDS-UPDRS III Axial Subscore (OFF DBS to Illumina 3D) | Baseline (OFF DBS) and after 45 minutes of Illumina 3D DBS
  Axial-related items of the MDS-UPDRS III, which includes items 3.1, 3.2, and 3.9-3.14. Each item is scored on a scale from 0 (normal) to 4 (severe), with the total possible score ranging from 0 to 32. A secondary outcome is the difference in MDS-UPDRS III Axial subscore from the OFF DBS condition (Baseline) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in QDG Mobility Score (SoC DBS to Illumina 3D) | After 45 minutes of Illumina 3D DBS and 45 minutes SoC DBS
  Quantitative Digitography (QDG) Mobility Score is a single score representing a participant's overall movement proficiency by combining performance across different aspects of movement including speed, frequency, amplitude, and rhythmicity measured using an engineered Keyduo QDG device during an alternating finger pressing and releasing with the index and middle finger. It is represented by a single value between 0 and 100 for each hand, where 100 represents ideal performance. A secondary outcome is the difference in QDG Mobility Score from the Standard of Care (SoC) DBS condition to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG mobility score will be used.
Change in QDG Tremor Severity Score (SoC DBS to Illumina 3D) | After 45 minutes of Illumina 3D DBS and 45 minutes SoC DBS
  A single score representing the proportion and amplitude of tremor-identified strikes using an engineered Keyduo QDG device. It is represented by a single value between 0 and 100, where 100 represents the worst tremor severity. A secondary outcome is the difference in QDG Mobility Score from the Standard of Care (SoC) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in QDG Percent Rest Tremor (SoC DBS to Illumina 3D) | After 45 minutes of Illumina 3D DBS and 45 minutes SoC DBS
  The proportion of tremor-identified strikes using an engineered Keyduo QDG device. Range from 0 to 100%. A secondary outcome is the difference in QDG Mobility Score from the Standard of Care (SoC) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in QDG Press Amplitude (SoC DBS to Illumina 3D) | After 45 minutes of Illumina 3D DBS and 45 minutes SoC DBS
  The average amplitude of strikes using an engineered Keyduo QDG device. Ranges from 0 to 14 mm. A secondary outcome is the difference in QDG Press Amplitude from the Standard of Care (SoC) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in QDG Press Amplitude Coefficient of Variation (SoC DBS to Illumina 3D) | After 45 minutes of Illumina 3D DBS and 45 minutes SoC DBS
  The coefficient of variation of press amplitude of strikes using an engineered Keyduo QDG device. A secondary outcome is the difference in QDG Press Amplitude Coefficient of Variation from the Standard of Care (SoC) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in QDG Interstrike Interval (SoC DBS to Illumina 3D) | After 45 minutes of Illumina 3D DBS and 45 minutes SoC DBS
  The interstrike-interval (i.e., the time it takes to complete one full press and release of the lever) of alternating tapping will be measured using an engineered Keyduo QDG device. The interstrike-interval is a time in milliseconds. A secondary outcome is the difference in QDG Interstrike Interval from the Standard of Care (SoC) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in QDG Release Slope (SoC DBS to Illumina 3D). | After 45 minutes of Illumina 3D DBS and 45 minutes SoC DBS
  The average speed of release using an engineered Keyduo QDG device. Units of cm/s. A secondary outcome is the difference in QDG Release Slope from the Standard of Care (SoC) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in QDG Press Speed (SoC DBS to Illumina 3D) | After 45 minutes of Illumina 3D DBS and 45 minutes SoC DBS
  The average speed of the press using an engineered Keyduo QDG device. Units of cm/s. A secondary outcome is the difference in QDG Press Speed from the Standard of Care (SoC) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in QDG Interstrike Interval Coefficient of Variation (SoC DBS to Illumina 3D) | After 45 minutes of Illumina 3D DBS and 45 minutes SoC DBS
  The variability of the interstrike-interval of alternating tapping, as quantified by the coefficient of variation, will be measured using an engineered Keyduo QDG device. A secondary outcome is the difference in QDG Interstrike Interval Coefficient of Variation from the Standard of Care (SoC) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in QDG Percent Freezing (SoC DBS to Illumina 3D) | After 45 minutes of Illumina 3D DBS and 45 minutes SoC DBS
  Proportion of freezing of finger tapping using a validated algorithm. Range from 0 to 100%. A secondary outcome is the difference in QDG Percent Freezingfrom the Standard of Care (SoC) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in Gait Speed (SoC DBS to Illumina 3D) | After 45 minutes of Illumina 3D DBS and 45 minutes SoC DBS
  The time it takes a person to walk a specified distance on level ground as measured by the GaitRite. Reported as m/s. A secondary outcome is the difference in Gait Speed from the Standard of Care (SoC) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in Gait Arrhythmicity (SoC DBS to Illumina 3D) | After 45 minutes of Illumina 3D DBS and 45 minutes SoC DBS
  Stride (gait cycle) time will be measured using the GaitRite. Gait arrhythmicity is defined as the mean stride time coefficient of variation (CV) of both legs. A greater stride time CV is indicative of less rhythmic gait/stepping. A secondary outcome is the difference in Gait Arrhythmicity from the Standard of Care (SoC) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in MDS-UPDRS III Total Score (SoC DBS to Illumina 3D) | After 45 minutes of Illumina 3D DBS and 45 minutes SoC DBS
  PD symptoms will be assessed clinically using the MDS-Unified Parkinson's Disease Rating Scale (UPDRS) Section III. This is a motor examination to evaluate speech, facial expression, tremor at rest, action or postural tremor of hands, rigidity, finger taps, hand movements, rapid alternating movement of hands, leg agility, arising from chair, posture, gait, freezing of gait, posture, body bradykinesia, and postural stability. Each item is scored on a scale from 0 (normal) to 4 (severe), with the total possible score ranging from 0 to 132. A secondary outcome is the difference in MDS-UPDRS III from the Standard of Care (SoC) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in MDS-UPDRS III Bradykinesia Subscore (SoC DBS to Illumina 3D) | After 45 minutes of Illumina 3D DBS and 45 minutes SoC DBS
  Bradykinesia-related items of the MDS-UPDRS III. Each item is scored on a scale from 0 (normal) to 4 (severe), with the total possible score ranging from 0 to 40.
  A secondary outcome is the difference in MDS-UPDRS III Bradykinesia subscore from the Standard of Care (SoC) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in MDS-UPDRS III Rigidity Subscore (SoC DBS to Illumina 3D | After 45 minutes of Illumina 3D DBS and 45 minutes SoC DBS
  Rigidity-related items of the MDS-UPDRS III. Each item is scored on a scale from 0 (normal) to 4 (severe), with the total possible score ranging from 0 to 20. A secondary outcome is the difference in MDS-UPDRS III Rigidity subscrore from the Standard of Care (SoC) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in MDS-UPDRS III Tremor Subscore (SoC DBS to Illumina 3D) | After 45 minutes of Illumina 3D DBS and 45 minutes SoC DBS
  Tremor-related items of the MDS-UPDRS III. Each item is scored on a scale from 0 (normal) to 4 (severe), with the total possible score ranging from 0 to 40. A secondary outcome is the difference in MDS-UPDRS III Tremor subscore from the Standard of Care (SoC) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used
Change in MDS-UPDRS III Axial Subscore (SoC DBS to Illumina 3D) | After 45 minutes of Illumina 3D DBS and 45 minutes SoC DBS
  Axial-related items of the MDS-UPDRS III. Each item is scored on a scale from 0 (normal) to 4 (severe), with the total possible score ranging from 0 to 32. A secondary outcome is the difference in MDS-UPDRS III Axial subscore from the Standard of Care (SoC) to Illumina 3D DBS. The Illumina 3D DBS amplitude condition with the highest QDG Mobility Score will be used

CONTACTS AND LOCATIONS:
Overall Officials: Helen Bronte-Stewart, MD, MSE, Principal Investigator — Stanford University
Locations (1):
- Stanford Neuroscience Health Clinic, Stanford, California, United States